CLINICAL TRIAL: NCT01396434
Title: A Non-interventional Study Of The Safety Of Pneumococcal 13-valent Conjugate Vaccine (Prevenar 13) In The Philippines: A Post Marketing Surveillance Study
Brief Title: Safety Surveillance of Pneumococcal 13-valent Conjugate Vaccine Among Filipinos
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1851076
Record Dates: First submitted 2011-06-22; First posted 2011-07-18 (Estimated); Results first posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-01

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prevenar 13 patients
  Interventions: Biological: Prevenar 13

INTERVENTIONS:
Biological: Prevenar 13 — Prevenar 13 vaccine as prescribed by the physician based on approved product indication
  Other Names: Pneumococcal 13-valent Conjugate Vaccine (13vPnC)

SUMMARY:
Prevenar 13 is safe for administration to Filipinos.

DETAILED DESCRIPTION:
Filipino patients prescribed and administered with the vaccine will be monitored for safety Patients prescribed with the vaccine who provides consent for inclusion to the study will be observed.

ELIGIBILITY:
Inclusion Criteria:

Patients prescribed with the vaccine

Exclusion Criteria:

Patients with hypersensitivity to the vaccine

Min Age: 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Filipino patients prescribed with the vaccine
Sampling Method: Non-Probability Sample
Enrollment: 3006 (Actual)
Dates: Start 2011-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (117):
- Philippines (117):
  - Private Clinic, Lipa City, Batangas
  - Private Clinic, Tagbilaran City, Bohol
  - Private Clinic, Malolos, Bulacan
  - Cebu Doctor University Hospital, Cebu, Cebu
  - Room 220 The Doctor's Hospital, Inc., Bacolod City, Negros Occidental
  - Private Clinic, San Carlos City, Negros Occidental
  - San Carlos Doctor's Hospital, San Carlos City, Negros Occidental
  - Victorias Commercial Center, Victorias City, Negros Occidental
  - Private Clinic, Dagupan, Pangasinan
  - Private Clinic, Mangaldan, Pangasinan
  - Private Clinic, Pozorrubio, Pangasinan
  - Private Clinic, Angeles City
  - Private Clinic, Antipolo City
  - Dr. Pablo O. Torre Memorial Medical Center, Bacolod City
  - Medical Arts Building, Bacolod City
  - Medical Plaza, Bacolod City
  - Private Clinic, Bacolod City
  - Riverside Medical Center, Bacolod City
  - Room 302 Medical Arts Building, Bacolod City
  - Room 311 Riverside Medical Arts Building, Bacolod City
  - Villanueva Laboratory and Clinics, Bacolod City
  - MCA Bauanan Children's Clinic, Batangas
  - Private Clinic, Batangas
  - Metropolitan Medical Center, Binondo, Manila
  - Private Clinic, Bocaue
  - 417, Bulacan
  - Clinica Tapia, Bulacan
  - Pediatric Doctor's Clinic, Bulacan
  - Private Clinic, Bulacan
  - St Vincent's Wellness Clinic, Bulacan
  - Room 11, Cagayan de Oro
  - Centralle Medical Diagnostics and Polyclinic, Caloocan
  - Private Clinic, Caloocan
  - Private Clinic, Candelaria
  - Blk 19 Lot 11, Capiz
  - Private Clinic, Cavite
  - Chong Hua Hospital, Cebu
  - Basement, Cebu City
  - Care and Cure Hub, Cebu City
  - Cebu Doctors University Hopsital, Cebu City
  - Chong Hua Hospital, Cebu City
  - PPG, Manila, Philippines, Cebu City
  - Private Clinic, Cebu City
  - Rm4A, Medical Arts Building, Cebu City
  - Room 302-A, Cebu City
  - Room 413 Medical Arts Building 2, Cebu City
  - Room 419 SPC Medical Specialty Center, Cebu City
  - Room 505A Chong Hua Medical Arts Building, Cebu City
  - Private Clinic, Dagupan
  - Community Health and Development Cooperative Hospital, Davao City
  - Health Science and Wellness Center, Davao City
  - Jesusa Complex, Davao City
  - Private Clinic, Davao City
  - San Pedro Hospital Inc., Davao City
  - San Pedro Hospital, Davao City
  - Private Clinic, Dipolog City
  - Private Clinic, Dumaguete
  - Room 117 Medical Arts Building, Dumaguete
  - Iligan Specialist Clinic, Iligan City
  - Private Clinic, Iloilo City
  - Private Clinic, Koronadal
  - Private Clinic, Laguna
  - Las Pinas Doctors Hospital, Las Piñas
  - Private Clinic, Legaspi
  - Private Clinic, Lipa City
  - Lucena United Doctors Hospital, Lucena City
  - Private Clinic, Lucena City
  - Private Clinic, Makati City
  - Archangel Raphael Pediatric Clinic, Malabon
  - Children's Clinic, Malabon
  - Malabon Medical Clinic, Malabon
  - Tumbicon Polycare, Malabon
  - Private Clinic, Malolos
  - Private Clinic, Mandaluyong
  - Metropolitan Medical Center, Manila
  - 1952, Manila
  - Children's Clinic, Manila
  - Chinese General Hospital, Manila
  - Private Clinic, Manila
  - Rm714B, Manila
  - Room 210, Metropolitan Medical Center, Manila
  - Room 706, Manila
  - Marikina Valley Medical Center, Marikina City
  - Centro Medical and Laboratory Clinic, Marikina City
  - Garcia General Hospital, Marikina City
  - Private Clinic, Marikina City
  - Room 605, Marikina City
  - Private Clinic, Negors Occidental
  - Private Clinic, Negros Occidental
  - Mabalacat Child Care Clinic, Pampanga
  - Private Clinic, Pangasinan
  - Maglana Villamor Clinic, Paranaque City
  - Paranaque Doctors Hospital, Paranaque City
  - Private Clinic, Pasig
  - Emil-Joanna General Hospital, Quezon
  - Private Clinic, Quezon
  - Philippine Heart Center, Quezon City
  - Friendly Care Clinic, Quezon City
  - Madrid Polyclinic, Quezon City
  - Maternity and Children's Clinic, Quezon City
  - Medical Specialist Clinic, Quezon City
  - Natividad Children's Clinic, Quezon City
  - Private Clinic, Quezon City
  - Room 11, Quezon City
  - World Citi Medical Center, Quezon City
  - Children'S Clinic, Rizal
  - Private Clinic, Rizal
  - Community General Hospital, San Pablo
  - Private Clinic, San Pablo
  - Chinese General Hospital and Medical Center, Santa Cruz, Manila
  - Private Clinic, South Luzon
  - Private Clinic, Tagbilaran City
  - Private Clinic, Tarlac City
  - Private Clinic, Urdaneta
  - Private Clinic, Valenzuela
  - Private Clinic, Zamboanga City
  - Room 331, Zamboanga City

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1851076&StudyName=Safety%20Surveillance%20of%20Pneumococcal%2013-valent%20Conjugate%20Vaccine%20Among%20Filipinos

RESULTS

PARTICIPANT FLOW:
Groups:
- 13vPnC (Prevenar 13), Cohort 1: Pneumococcal 13-valent conjugate vaccine (13vPnC) as prescribed by the physician based on approved product indication for infants and children 6 weeks through 5 years of age.
- 13vPnC (Prevenar 13), Cohort 2: 13vPnC as prescribed by the physician based on approved product indication for adults 50 years and older.
- 13vPnC (Prevenar 13), Cohort 3: 13vPnC as prescribed by the physician based on approved product indication. These participants may have had incorrect documentation of their 13vPnC vaccine date(s) and were neither included in the 6 weeks through 5 years of age nor 50 years and older indication group.
Period: Overall Study
Arm/Group | 13vPnC (Prevenar 13), Cohort 1 | 13vPnC (Prevenar 13), Cohort 2 | 13vPnC (Prevenar 13), Cohort 3
Started | 2817 | 175 | 14
Completed | 2806 | 175 | 14
Not Completed | 11 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Other | 10 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of 13vPnC.
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC (Prevenar 13), Cohort 1 | 13vPnC (Prevenar 13), Cohort 2 | 13vPnC (Prevenar 13), Cohort 3 | Total
Number analyzed (Participants) | 2817 | 175 | 14 | 3006
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age at enrollment (years) | 0.5 (0.94) | 65.1 (10.60) | 0.7 (1.54) | 4.3 (15.37)
Gender [Count of Participants; unit: Participants]
  Female | 1402 | 115 | 6 | 1523
  Male | 1415 | 60 | 8 | 1483
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 2783 | 175 | 14 | 2972
  Other | 24 | 0 | 0 | 24
  White | 8 | 0 | 0 | 8
  Black | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: All observed or volunteered AEs and SAEs regardless of treatment group or suspected causal relationship to 13vPnC were reported. An AE was any untoward medical occurrence in a participant who received 13vPnC. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-SAEs.
Time Frame: Baseline through and including 28 calendar days after the last administration of study vaccine within the observation period
Population: Participants who received at least 1 dose of 13vPnC.
Measure: Number; unit: participants
Arm/Group | 13vPnC (Prevenar 13), Cohort 1 | 13vPnC (Prevenar 13), Cohort 2 | 13vPnC (Prevenar 13), Cohort 3
Number analyzed (Participants) | 2817 | 175 | 14
participants
  AEs | 68 | 5 | 0
  SAEs | 1 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | 13vPnC (Prevenar 13), Cohort 1 | 13vPnC (Prevenar 13), Cohort 2 | 13vPnC (Prevenar 13), Cohort 3
Serious Adverse Events (participants affected / at risk) | 1/2817 | 0/175 | 0/14
Other Adverse Events (participants affected / at risk) | 68/2817 | 5/175 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 13vPnC (Prevenar 13), Cohort 1 (N=2817) | 13vPnC (Prevenar 13), Cohort 2 (N=175) | 13vPnC (Prevenar 13), Cohort 3 (N=14)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 13vPnC (Prevenar 13), Cohort 1 (N=2817) | 13vPnC (Prevenar 13), Cohort 2 (N=175) | 13vPnC (Prevenar 13), Cohort 3 (N=14)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 38 (38) | 2 (2) | 0 (0)
Injection site pain (General disorders) | 3 (3) | 0 (0) | 0 (0)
Swelling (General disorders) | 2 (2) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Crying (General disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Viral rash (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Amoebiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The use of 13vPnC was based on the investigator's clinical judgment and was assumed to be consistent with the product's approved label.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less